CLINICAL TRIAL: NCT02344043
Title: Cerebral Oxygenation and Neurological Outcomes FOllowing CriticAL Illness
Acronym: CONFOCAL
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Gordon Boyd, Assistant Professor, Queen's University
Other Study IDs: DMED-1662-13
Record Dates: First submitted 2015-01-08; First posted 2015-01-22 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Critical Illness; Sepsis; Delirium; Respiratory Failure
MeSH Terms: conditions — Critical Illness; Sepsis; Delirium; Respiratory Insufficiency | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critical illness: This prospective cohort of critically ill patients will have brain tissue oxygen levels recorded for 24 hours after admission with near infrared spectroscopy.
  Interventions: Device: Near infrared spectroscopy

INTERVENTIONS:
Device: Near infrared spectroscopy — This device uses near infrared spectroscopy to measure tissue oxygen levels (0-100%). The sensors are placed on the subjects' forehead to measure brain tissue oxygenation

SUMMARY:
Purpose of the Study Critical illness requiring life support affects over 150 000 people in Ontario every year. With aggressive support, the number of people who die from critical illness is decreasing. However, people who survive often have neurological problems. These neurological problems often include difficulties with memory, concentration, and attention. These problems are associated with poor quality of life among survivors of critical illness. The aim of this study is to identify the factors that contribute to these neurological deficits. Specifically, the investigators are testing whether changes in oxygen delivery to the brain during critical illness are related to both short- and long-term neurological complications.

Procedures involved in the Research When patients are diagnosed with a critical illness such as shock or respiratory failure, they are treated with intravenous fluids, medications to raise their blood pressure, and can be placed on a ventilator to assist with their breathing. They are observed in an intensive care unit (ICU). This research protocol does NOT interfere with the normal treatment of patients with critical illness. The procedure involved in this research protocol requires the placement of two stickers to either side of the patient's forehead, and information about oxygen delivery to the brain will be recorded. When the patient has recovered from the critical illness, they will be asked to perform several neurological tests. Some of these tests will be done with a pencil and paper, while others will use a robotic device to test arm movements, reaction time, and concentration.

Potential Harms, Risks or Discomforts:

This research study involves the placement of a sticker sensor to either side of the forehead. Rarely, patients may develop a rash to these electrodes. The investigators monitor patients very carefully for rashes, and if a rash is to occur, the sticker sensor will be removed. With regards to the neurological testing, rarely patients can have some mild muscle stiffness after moving their arms in the robot. The investigators do not expect any other further harms, risks, or discomforts.

DETAILED DESCRIPTION:
A detailed protocol is currently under review for funding at Physician Services Incorporated, and can be included pending decision.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients defined as having either:

  1. Respiratory failure: Defined as invasive mechanical ventilation for a predicted duration of >24 hours, or:
  2. Shock: Defined as being on one of the following agents:
* norepinephrine (>5 mcg/min) IV
* epinephrine (at any dose)
* vasopressin (in combination with another pressor)
* milrinone (in combination with another pressor)

Exclusion Criteria:

* expected survival <24 hours
* history of cognitive dysfunction
* unable to participate in follow up testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is recruiting critically ill patients admitted to the 33-bed medical/surgical intensive care unit at an academic medical centre.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Delirium | Proportion of ICU stay spent delirious. The average ICU stay is 7 days at our institution, however, some patients may stay much longer. We will perform delirium screening to a maximum of 30 days after ICU admission.
  The CAM-ICU and ICDSC are used to screen for delirium in critically ill patients. On the basis of these two validated screening tools, patients will be categorized as either comatose, delirious, or intact. The percentage of ICU stay that the participant spends delirious is the primary outcome measure.

SECONDARY OUTCOMES:
Neurocognitive performance on KINARM tasks | 3 and 12 months
  The KINARM is a robotic device that provides quantitative metrics of the neurocognitive control of upper arm movements.
Neurocognitive performance on the RBANS | 3 and 12 months
  The RBANS is the repeatable battery for the assessment of neuropsychological status
Correlation between brain tissue oxygenation and physiological parameters | First 24 hours of admission
  We will use correlation coefficients to describe the relationship between brain tissue oxygenation and physiological parameters recorded during the first 24 hours of critical illness.

CONTACTS AND LOCATIONS:
Overall Officials: John G Boyd, MD, PhD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will publish our data in a peer reviewed scientific journal

REFERENCES:
- [Derived] Khan JM, Shore A, Lee KFH, Wood MD, Maslove DM, Hunt M, Georgescu I, Muscedere J, Boyd JG. Cerebral autoregulation-based mean arterial pressure targets and delirium in critically ill adults without brain injury: a retrospective cohort study. Can J Anaesth. 2024 Jan;71(1):107-117. doi: 10.1007/s12630-023-02609-w. Epub 2023 Nov 6. PMID 37932650
- [Derived] Wood MD, Jacobson JA, Maslove DM, Muscedere JG, Boyd JG; Cerebral Oxygenation and Neurological Outcomes Following Critical Illness (CONFOCAL) Research Group. The physiological determinants of near-infrared spectroscopy-derived regional cerebral oxygenation in critically ill adults. Intensive Care Med Exp. 2019 May 2;7(1):23. doi: 10.1186/s40635-019-0247-0. PMID 31049754
- [Derived] Wood MD, Maslove DM, Muscedere J, Scott SH, Boyd JG; Canadian Critical Care Trials Group. Robotic technology provides objective and quantifiable metrics of neurocognitive functioning in survivors of critical illness:A feasibility study. J Crit Care. 2018 Dec;48:228-236. doi: 10.1016/j.jcrc.2018.09.011. Epub 2018 Sep 12. PMID 30243203
- [Derived] Cerebral Oxygenation and Neurological Outcomes Following Critical Illness (CONFOCAL) Research Group; Canadian Critical Care Trials Group; Wood MD, Maslove DM, Muscedere JG, Day AG, Gordon Boyd J. Low brain tissue oxygenation contributes to the development of delirium in critically ill patients: A prospective observational study. J Crit Care. 2017 Oct;41:289-295. doi: 10.1016/j.jcrc.2017.06.009. Epub 2017 Jun 15. PMID 28668768